CLINICAL TRIAL: NCT02151890
Title: Pregnancy After Stem Cell Transplantation in Premature Ovarian Failure (POF)
Brief Title: Pregnancy After Stem Cell Transplantation in Premature Ovarian Failure
Acronym: POF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Edessy Mahmoud, Professor, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Al Azhar University; POF women (Registry Identifier: Al Azhar U); Stem cell transplantation (Registry Identifier: Al Azhar University)
Record Dates: First submitted 2014-05-22; First posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Premature Ovarian Failure
Keywords: POF; ESS; stem cell
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laparoscopic Stem Cell Transplantation. (Experimental): Out of 112 high risk patients for POF diagnosis was established in 10 cases. Endometrial fractional biopsy was taken, stained with H&E stain and by IH staining by stem cell marker OCT4. Immunohistochemical expression of stem cell marker OCT4 was evaluated before and after transplantation according to Edessy Stem Cell Scoring (ESS)Laparoscopic injected of stem cell Sample in the ovaries.. Participants were followed up monthly for a period of six months by hormonal (FSH, LH and E2), clinical (resuming menstruation), US (folliculometry), histopathological (HP), and IH expression of stem cell marker OCT4 of the endometrial biopsy (stem cell positivity according to ESS) outcome.
  Interventions: Biological: Stem Cell

INTERVENTIONS:
Biological: Stem Cell — Out of 112 high risk patients for POF diagnosis was established in 10 cases. Endometrial fractional biopsy was taken, stained with H&E stain and by Immunohistochemical (IH) staining by stem cell marker OCT4. IH expression of stem cell was evaluated before and after transplantation according to Edessy Stem Cell Scoring (ESS). After laparoscopic injection of stem cell sample in the ovaries, participants were followed up monthly for a period of one year by hormonal (FSH, LH and E2), clinical (resuming menstruation and pregnancy), US (folliculometry), histopathological (HP), and IH expression of stem cell (stem cell positivity and scoring according to ESS).
  Other Names: - Edessy Stem cell Score.; - Laparoscopic stem cell transplantation.; - Hormonal Analysis; - Ultrasonic evaluation

SUMMARY:
Out of 112 high risk patients for Premature Ovarian Failure (POF), diagnosis was established in 10 cases.

ESS cut off point for menstruation and pregnancy was 6.

DETAILED DESCRIPTION:
Out of 112 high risk patients for POF, diagnosis was established in 10 cases. Endometrial fractional biopsy was taken, stained with H&E stain and by immubohistchemical (IH) staining by stem cell marker OCT4. IH expression of stem cell marker OCT4 was evaluated before and after transplantation according to Edessy Stem Cell Score (ESS).

After laparoscopic injection of stem cell sample in the ovaries, participants were followed up monthly for a period of one year by hormonal (FSH, LH and E2), clinical (resuming menstruation), US (folliculometry), histopathological (HP), and IH expression of stem cell (stem cell positivity and scoring according to ESS).

These cases were of ESS 5 and 6.

ELIGIBILITY:
Inclusion Criteria:

* Post-menarche female less than 40 years old.
* Normal karyotyping female.
* Primary ovarian failure females
* Follicle-stimulating hormone (FSH) more than or equal to 20 IU/L.
* Agree to sign the designed consent for the study.

Exclusion Criteria:

* Autoimmune diseases.
* Breast cancer, ovarian cancer.
* Hypersensitivity to any Gonadotropin-releasing hormone (GnRH) analogs.
* Those with major medical problems such as malignancy, hepatitis, etc.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Pregnancy | 104 weeks
  Hormonal analysis

SECONDARY OUTCOMES:
Menstruation | 104 weeks
  Clinical

OTHER OUTCOMES:
Ovulation | 104 weeks
  Ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Edessy, Professor, Principal Investigator — Al-Azhar University; Hala N Hosni, Professor, Study Chair — Cairo University; Yehia Wafa, Professor, Study Chair — Al-Azhar University; Yousef Shady, MD, Study Chair — Al-Azhar University; Sayed Bakri, MD, Study Chair — Al-Azhar University; Medhat Kamel, Msc, Study Chair — Al-Azhar University
Locations (1):
- Al Azhar University, Cairo, Cairo Governorate, Egypt